CLINICAL TRIAL: NCT03723317
Title: Associated Balance of Risk Score - Comprehensive Complication Index for the Prediction of Long-term Survival After Liver Transplantation
Brief Title: Associated Balance of Risk Score - Comprehensive Complication Index for the Prediction of Post-transplant Survival
Status: Completed | Type: Observational
Sponsor: European Hepatocellular Cancer Liver Transplant Group (Other)
Responsible Party: Sponsor
Other Study IDs: #0003
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Liver Cirrhosis; Liver Failure; Liver Diseases; Transplant Failure
MeSH Terms: conditions — Liver Cirrhosis; Liver Failure; Liver Diseases | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training liver transplantation: Patients consecutively transplanted in four European collaborative LT Centres (Ancona, Brussels, Rome Sapienza, and Padua) (N=1,262)
  Interventions: Procedure: Liver transplantation
- Validation liver transplantation: Patients consecutively transplanted in the Karolinska Institute (N=520)
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — First deceased-donor liver transplantation

SUMMARY:
In recent years, several scoring systems have been developed aimed at predicting early post-LT graft function. However, many of them showed poor efficacy when long-term survivals were tested. Moreover, the necessity to find an easy-to-use score represents another obstacle, with several scores composed by numerous, difficult to find, variables. Recently, the pre-LT Balance of Risk (BAR) and the post-LT Comprehensive Complication Index (CCI) have been created, but their external validation and integration in this setting is lacking.

This study aims at constructing an easy-to-use score system based on the combination of a small number of pre- and immediately post-liver transplant (LT) independent variables, in order to accurately predict long-term graft survival after LT.

DETAILED DESCRIPTION:
In the last years, several scoring systems have been developed with the intent to predict waiting-list mortality or early allograft dysfunction (EAD) after liver transplantation (LT). The Model for End-stage Liver Disease (MELD) is recognised as the most accurate liver allograft allocation model by prioritising patients according to the severity of their disease. However, several studies showed that MELD alone failed to predict early and late post-transplant clinical course. Consequently, other scoring systems based on pre-LT or post-LT variables have been developed, with the intent to identify high-risk cases for death, graft loss or re-transplantation (re-LT). Among them, two pre-LT scores, namely the D-MELD and Balance of Risk (BAR), showed to well predict early post-LT survival. Similarly, some post-LT scores were able to estimate EAD, and, thereby, to predict the probabilities of early re-LT and patient death. Interestingly, all of these scores, especially those based on pre-LT variables, resulted in a scarce prediction of long-term (five-year) survivals.

Recently, the Comprehensive Complication Index (CCI) has been developed in order to better capture complication rates after surgery. Some reports reported its excellent prognostic ability in different fields. However, up to now, no studies investigated the role of CCI concerning long-term prognostication of graft loss in LT.

This study aims at constructing an easy-to-use score system based on the combination of a small number of pre- and immediately post-LT independent variables, in order to accurately predict five-year post-LT graft survival. Both external and internal validations of the score were performed.

ELIGIBILITY:
Inclusion Criteria:

* First transplant
* adult (>18 years)

Exclusion Criteria:

* living donation
* re-transplant
* combined transplant
* domino transplant
* paediatric transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients transplanted for any liver pathology undergoing a first transplant.
Sampling Method: Probability Sample
Enrollment: 1782 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Five-year post-transplant graft survival | 5 years
  Number of participants experiencing a graft loss for any reason

SECONDARY OUTCOMES:
Re-transplant rate | 5 years
  Number of participants experiencing a re-transplant for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Quirino Lai, MD PhD, Principal Investigator — UCL Brussels
Locations (1):
- UCL, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai Q, Melandro F, Nowak G, Nicolini D, Iesari S, Fasolo E, Mennini G, Romano A, Mocchegiani F, Ackenine K, Polacco M, Marinelli L, Ciccarelli O, Zanus G, Vivarelli M, Cillo U, Rossi M, Ericzon BG, Lerut J. The role of the comprehensive complication index for the prediction of survival after liver transplantation. Updates Surg. 2021 Feb;73(1):209-221. doi: 10.1007/s13304-020-00878-4. Epub 2020 Sep 6. PMID 32892294